CLINICAL TRIAL: NCT04845152
Title: Prevalence of Migraine Disease in Electrohypersensitive Patients
Brief Title: Migraine in Electrohypersensitive Patients
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0250
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Headache; Migraine
Keywords: Electrohypersensitivity
MeSH Terms: conditions — Headache; Migraine Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators propose here by the use of the French version of the migraine disease screening questionnaire (ID Migraine ™) to study the prevalence of migraine disease in a population of electrohypersensitive patients

ELIGIBILITY:
Inclusion criteria:

* Informed Consent
* 18 years or older at the time of informed consent

With all these criteria :

* the perception by the subjects of various non-specific functional symptoms
* the absence of clinical and biological evidence to explain the symptoms
* the attribution by the subjects themselves of these symptoms to exposure to electromagnetic fields, which are themselves diverse
* the symptoms are chronic (more than 3 months)
* the symptoms appear during an exposure to a source of electromagnetic radiation and cease after the exposure is stopped
* the symptoms are reproducible

Exclusion criteria:

- age under 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: An adult declaring himself electrohypersensitive
Sampling Method: Non-Probability Sample
Enrollment: 317 (Actual)
Dates: Start 2021-04-30 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Possible migraine attack | 12 months
  With the number of positive response to the French version of the migraine disease screening questionnaire, we are looking for the patients declaring themselves electrohypersensitive if they have had headaches in the last 12 months with characteristics that could evoke a migraine attack.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric GRECO, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC